CLINICAL TRIAL: NCT03729622
Title: A Pilot Randomised Controlled Trial of the Effect of a Diet Low in Poorly Digested Carbohydrates on Gastrointestinal Form and Symptoms in Irritable Bowel Syndrome Patients
Brief Title: Carbohydrate Reduction and Impact on Gastrointestinal System
Acronym: CRAIGS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15081
Record Dates: First submitted 2017-08-18; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-11

CONDITIONS: Irritable Bowel Syndrome
Keywords: FODMAPs; Low FODMAP Diet
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Intervention (Active Comparator): Participants in this arm will receive an immediate low FODMAP dietary intervention on their second visit after they have been screened, consented and enrolled during visit 1.
  Interventions: Other: Low FODMAP Diet
- Delayed Intervention (Placebo Comparator): Participants in this arm will receive a delayed Low FODMAP dietary intervention during their third visit after they have been been screened, consented and enrolled during visit 1.
  Interventions: Other: Low FODMAP Diet

INTERVENTIONS:
Other: Low FODMAP Diet — Both arms will receive the intervention but at different time points.

SUMMARY:
Title :

A pilot single blind randomised controlled trial of the effect of a diet low in poorly digested carbohydrates on gastrointestinal form and symptoms in irritable bowel syndrome patients

Acronym: CRAIGS

Short title: Carbohydrate reduction and impact on gastrointestinal system Chief Investigator: Prof Robin Spiller

Objectives:

The purpose of this study is to:

* Investigate the proportion of patients with Irritable Bowel Syndrome who report moderate or substantial improvement in their symptoms after 2 weeks of following a diet low in Fermentable Oligo-Di-Monosaccharides and Polyols (FODMAPs) compared to patients who are on their habitual diet.
* Determine the difference in colonic volume of IBS patients receiving immediate low FODMAP dietary intervention after 2 weeks compared to patients who are not on the diet (delayed dietary intervention).
* Investigate the changes in self-reported food intolerance that occurs before dietary intervention.

Trial Configuration:

2-arm, parallel group, randomised, controlled trial

Setting :

Research clinic within NIHR Biomedical Research Unit, Secondary care

DETAILED DESCRIPTION:
TRIAL / STUDY OBJECTIVES AND PURPOSE

The trial aims to investigate the effect of a diet low in FODMAPs on colonic morphology as well as in improving symptoms of irritable bowel syndrome (IBS).

This mechanistic information, along with the clinical data, will allow planning of larger, multi-centre studies of the low FODMAP diet in similar patients.

HYPOTHESES

* Patients on a low FODMAP diet for 2 weeks will have a decreased fasting colonic volume measured by Magnetic Resonance Imaging (MRI) compared to participants who have not started the diet.
* Patients with IBS are more likely to report a clinically important improvement in symptoms following the low FODMAP diet (immediate intervention) compared to those on their habitual diet (delayed intervention).

PRIMARY OBJECTIVE • To compare the proportion of IBS patients reporting a clinically important improvement in symptoms following a low FODMAP diet for 2 weeks against IBS patients who are on their habitual diet.

SECONDARY OBJECTIVES

• Determine the difference in fasting colonic volume of IBS patients receiving low FODMAP dietary intervention after 2 weeks compared to those on habitual diet.

TRIAL DESIGN

This will be a pilot single-blind, randomised, controlled trial (RCT). Since some activity will take place on the University of Nottingham this will be a multi-centre study.

All participants will receive advice from a dietitian on the low FODMAP diet. They will be randomised to one of two parallel treatment arms:

1. Low FODMAP dietary advice (immediate intervention)
2. Habitual diet (control - delayed intervention )

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above
* Able to give informed consent
* Previous Diagnosis of IBS by medical practitioner
* Meeting ROME III criteria for IBS
* Investigations showing negative tissue transglutaminase (tTG) IgA antibodies
* Full blood count test does not indicate Anaemia

Exclusion Criteria:

* Inclusion

  * Aged 18 and above
  * Able to give informed consent
  * Previous Diagnosis of IBS by medical practitioner
  * Meeting ROME III criteria for IBS
  * Investigations showing negative tissue transglutaminase (tTG) IgA antibodies
  * Full blood count test does not indicate Anaemia

Exclusion

* Children (<18 years)
* History declared by the candidate of pre-existing gastrointestinal disorder, including but not limited to:

  * Inflammatory Bowel Disease
  * Coeliac Disease
  * Pancreatitis
  * Gallstone disease (biliary colic, cholecystitis)
  * Diverticulitis
  * Cancer of the gastrointestinal tract
* Reported history of previous resection of any part of the gastrointestinal tract other than appendix or gallbladder
* Intestinal stoma
* Limited understanding of English
* Pregnancy declared by the candidate
* Red flag symptoms such as rectal bleeding, family history of bowel or ovarian cancer, a change in bowel habit to looser and/or more frequent stools persisting for more than six weeks in a person aged over 60 years.
* Investigations showing positive tissue transglutaminase (tTG) IgA antibodies
* Anaemia confirmed by full blood count test
* Habitual use of opiate analgesics likely to alter bowel function e.g. morphine
* Use of antibiotics in the preceding four weeks other than for treatment of index infection.
* Any condition where the candidate is likely to require a course of antibiotics in the next 3 months e.g. severe chronic respiratory disease, recurrent urinary tract infection, lower limb ulceration
* Inability to complete the symptom questionnaires e.g. cognitive dysfunction limiting memory and understanding
* Anyone who in the opinion of the investigator is unlikely to be able to comply with the protocol e.g. chaotic lifestyle related to substance abuse
* Dietary practice not compatible with safe implementation of the trial diet e.g.veganism
* Medical reasons for pre-existing controlled diet that cannot be safely randomised e.g. end-stage kidney disease, diabetes
* Participants taking prebiotic/probiotic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Adequate symptom relief between cases and controls | Assessed in cases on their last day of the intervention (2 weeks after dietary change). Assessed in controls before they began their intervention (between 1-2 weeks before dietary changes)
  Adequate symptom relief assessed by questionnaire after intervention in cases and before intervention in cases

SECONDARY OUTCOMES:
Changes in colonic volume between cases and controls from baseline | Measured : i) baseline (day 0), ii) last day of intervention (cases) (2 weeks after dietary change), iii) before intervention (2 weeks before dietary advice)
  A change in colonic volume measured in milliliters (ml) from baseline and after intervention in cases. This will compared with a change in colonic volume from baseline and before intervention in controls.
Changes in fermentation between cases and controls | Measured : i) baseline (day 0), ii) last day of intervention (cases) (2 weeks after dietary change), iii) before intervention (2 weeks before dietary advice)
  A change in breath hydrogen concentration measured in parts per million (ppm) from: baseline and after intervention (cases) ii) from baseline and before intervention (controls)

CONTACTS AND LOCATIONS:
Overall Officials: Robin Spiller, MD,FRCP, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham Digestive Diseases Centre, Nottingham, Nottinghamshire, United Kingdom